CLINICAL TRIAL: NCT01665703
Title: LCCC 1213: Defining Molecular and Functional Imaging Correlates of Renal Cell Carcinoma Biological Features
Brief Title: Imaging Correlates of Renal Cell Carcinoma Biological Features
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC1213
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Renal Cell Carcinoma
Keywords: [18F]; Fluorodeoxyglucose Positron Emission Tomography-Magnetic Resonance Imaging; FDG-PET-MRI; Renal Cell Carcinoma; Pilot Study; LCCC 1213; UNC Lineberger
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FDG PET/MR (Experimental): Participents will undergo a gadolinium enhanced FDG PET/MR study.
  Interventions: Procedure: FDG PET/MR

INTERVENTIONS:
Procedure: FDG PET/MR — Patients will be asked to undergo a voluntary gadolinium enhanced MRI with simultaneous acquisition of FDG-PET uptake within 4 weeks prior to surgery.
  Other Names: Fluorodeoxyglucose Positron Emission Tomography MRI

SUMMARY:
This pilot study is designed to evaluate imaging parameters indicative of underlying tumor biology. Patients with large renal masses (>3 cm, or at the discretion of the investigator) who are planning to undergo nephrectomy will be identified, and recruited to undergo a contrast-enhanced magnetic resonance-Fluorodeoxyglucose-positron emission tomography (MR-FDG-PET) scan.

DETAILED DESCRIPTION:
This pilot study is designed to evaluate imaging parameters indicative of underlying tumor biology. Patients with large renal masses (>3 cm, or at the discretion of the investigator) who are planning to undergo nephrectomy will be identified, and recruited to undergo a contrast-enhanced magnetic resonance-Fluorodeoxyglucose-positron emission tomography (MR-FDG-PET) scan. Samples collected from their tumor after it is removed will undergo a variety of laboratory tests, including biomarker assessments and genotyping. By examining primary renal masses via a combination of MR and FDG-PET functional imaging in concert with tissue based tests, areas of hypermetabolism and hypervascularization will be evaluated as features of HIF activation or tumor subtype.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age (no upper age limit)
* Informed consent obtained and signed
* Clinically suspected RCC based on imaging performed prior to enrollment
* Planned nephrectomy schedule that can accommodate a MR-FDG-PET scan within 4 weeks prior to surgery
* Willing to undergo gadolinium enhanced MRI with simultaneous acquisition of FDG-PET uptake by the tumor within 4 weeks prior to nephrectomy
* Willing to consent for genetic and proteomic analysis of tumor and germline nucleic acids
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to FDG-PET-MRI
* Breast feeding women cannot do so for 24 hours after FDG injection
* Patient is willing to fast for 4 hours, including avoiding any sugar-containing drinks.
* Patient is willing to drink at least 32 ounces of water (or other no-sugar-containing fluids) within 4 hours prior to arriving for scans.

Exclusion Criteria:

* History of severe reaction to gadolinium-enhanced MRI
* Poorly controlled diabetes mellitus
* Inability to tolerate PET and/or MRI
* Presence of pacemaker or intracranial aneurysm clip
* GFR < 30mL/min as measured via Cockcroft-Gault equation
* Inability to lie flat for >1 hour
* Pregnant female
* History of a prior malignancy within past 5 years are excluded unless they have been disease free for 3 or more years or unless they have a completely resected non-melanoma skin cancer, low risk prostate cancer, or other low risk tumor history at the discretion of the investigator.
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-08; Primary Completion 2014-11 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of FDG-PET-MRI making useful measurements that might be then used to globally assess tumor biological features | 4 weeks
  This is a feasibility study. Feasibility will be determined by the quality of the FDG-PET-MRI measurements. That is, the measurements represent what the investigators hope they are measuring. With 10 of 10, the 100% rate has an exact 95% confidence interval of 69% to 100%. The interval width, representing a measure of precision, is 31%. The tumor biological features that will be assessed include genetic analyses performed for commonly mutated genes in kidney cancer (VHL, PBRM1, SETD2, HIF1, UTX, MLL2) and protein expression analyses performed on HIF1 and HIF2 protein expression using standard immunohistochemistry. These genetic and protein expression analyses will be performed on tissue samples collected within four weeks of imaging from tissue removed via nephrectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Lin, PhD, Principal Investigator — University of North Carolina
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Lineberger Comprehensive Cancer Center website — http://unclineberger.org/
- See also: National Cancer Institute (NCI) website — http://www.cancer.gov/